CLINICAL TRIAL: NCT01199952
Title: A Randomized Controlled Trial: Contraceptive Counseling After an Abortion
Brief Title: RCT: Can a Single Counseling Phone Call Improve Contraception After an Abortion?
Acronym: PPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RCT 10-01978
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-08

CONDITIONS: Contraception
Keywords: contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control group will not receive a counseling phone call one month after enrollment.
- Intervention (Experimental): Intervention arm receives a counseling phone call 3 to 4 weeks after enrollment. The call is from a health educator intended to assist with contraception.
  Interventions: Behavioral: Treatment group: receives counseling phone call intervention

INTERVENTIONS:
Behavioral: Treatment group: receives counseling phone call intervention — Subjects in the treatment arm will receive a phone call from a health educator to assist with contraception, 3 to 4 weeks after enrollment.
  Arms: Intervention

SUMMARY:
Hypothesis: Use of an effective contraceptive six weeks after abortion will be higher in the treatment group than in the control group.

Primary Aim ·To determine use of an effective contraceptive method six weeks after abortion in women who choose combined hormonal contraception (CHC) and who receive a three-week educational phone call as compared to women who do not receive the intervention.

Secondary Aims

* To describe the most common concerns and logistical problems women experience with initiating and adhering to CHC after abortion.
* To describe the concerns that lead to discontinuation or method change. *To assess feasibility of conducting a follow-up telephone call in this population This is a randomized, controlled trial to assess the effect of a three-week follow-up phone call in women who choose combined hormonal contraception on the day of their abortion at the San Francisco General Hospital Women's Options Center. Subjects randomized to the treatment group will receive an interventional phone call three weeks after their abortion; participants randomized to the control group will not receive the call. All subjects will receive a follow-up call six weeks after their abortion to assess and compare method use between the two groups. Calls will be made at three- and six-weeks post abortion in order to give subjects enough time to initiate CHC and to assess continuation into the second month of the method. Data will be collected at baseline, during the intervention for the treatment group and during the final follow-up call for both groups. The primary outcome is use of an effective contraceptive six weeks after abortion.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 15 who choose pill, patch or ring to begin after their abortion
* Women able and willing to be contacted by phone for up to 2 months after enrollment

Exclusion Criteria:

* Women who do not speak and read English or Spanish

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2011-03-21 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jody Steinauer, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were recruited at the county hospital abortion clinic from 3/21/2011 to 5/25/2012.
  Follow up phone calls were conducted 6 week and 6 months after enrollment, with the final follow-up completed 1/2/2013.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 103 | 104
Completed | 51 | 59
Not Completed | 52 | 45

BASELINE CHARACTERISTICS:
Population: The number of baseline participants matches the Participant Flow, n=207
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 103 | 104 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (4.9) | 24.4 (6.2) | 24.8 (6.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  only female in study | 103 | 104 | 207
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 11 | 19 | 30
  Race: African-American | 29 | 37 | 66
  Race: Hispanic | 36 | 22 | 58
  Race: Native American/Eskimo | 2 | 0 | 2
  Race: Native Hawaiian/Pacific Islander | 3 | 2 | 5
  Race: White | 18 | 18 | 36
  Race: Other | 1 | 3 | 4
  Race: Unknown | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Using an Effective Contraceptive Method 6 Weeks After Abortion
Description: To determine use of an effective contraceptive method six weeks after abortion in women who choose combined hormonal contraception (CHC) and who receive a three-week educational phone call as compared to women who do not receive the intervention.
Time Frame: 6 weeks after abortion procedure
Population: study sample is female only since study is birth control selected following surgical abortion
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 103 | 104
Participants | 55 | 55

2. Secondary Outcome: Reasons for Discontinuation of Contraception
Description: To describe the most common concerns and logistical problems women experience with initiating and adhering to CHC after abortion.
  To describe the concerns that lead to discontinuation or method change.
  To assess feasibility of conducting a follow-up telephone call in this population
Time Frame: 6 weeks after abortion procedure
Population: number who responded to 6 week follow-up contact responses to outcome measures were not mutually exclusive, and therefore will not add up to the total number of participants who responded to the six week survey/contact.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 69 | 75
Participants
  Stopped having sex | 14 | 11
  worried wouldn't be able to get pregnant | 7 | 6
  Couldn't afford it | 3 | 5
  Couldn't get more | 7 | 8
  My partner wanted me to stop using it | 2 | 2
  My doctor told me to stop | 1 | 1
  My friends thought that I should stop | 2 | 1
  Other reason | 18 | 15
  No other reason | 23 | 23

ADVERSE EVENTS:
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/104
Other Adverse Events (participants affected / at risk) | 0/103 | 0/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No